CLINICAL TRIAL: NCT04832737
Title: Could a Strength- Based Treatment Improve Self-management in Adults With Attention Deficit Hyperactivity Disorder
Brief Title: Strength-based Treatment Approach for Adults With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Huddersfield (Other)
Responsible Party: Principal Investigator, Rebecca Champ, Principal Investigator, University of Huddersfield
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC001
Record Dates: First submitted 2021-03-29; First posted 2021-04-06 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: This is a wait list control study design with pre-, within, and post-treatment measures. A rolling entry of participants will be conducted, where once individuals have been screened their entry into the study will begin. A maximum of 30 adults aged 18+ with a confirmed diagnosis of ADHD will be allocated using block randomisation to the SDT theory-based model or wait list over a 12-week period. Following the 12-week wait, the wait list group will also be enrolled in the SDT theory-based model. This ensures all participants receive the opportunity to experience the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): SDT theory-based psychotherapeutic treatment model
  Interventions: Behavioral: ADDapt Ability Framework
- Control (No Intervention): Wait List

INTERVENTIONS:
Behavioral: ADDapt Ability Framework — 12 week individual therapeutic coaching intervention
  Arms: Intervention

SUMMARY:
The aim of the research is to develop a treatment program with positive self-awareness and self-determination outcomes for adults with Attention Deficit Hyperactivity Disorder (ADHD). Current treatments are based in a characterisation of ADHD oriented on deficits impairing everyday functioning, with primary goals of symptom control and reduction. However, treatment approaches are not standardised and only evidence short-term effectiveness. This project proposes an alternative approach to understanding ADHD behaviours, supported by Self Determination Theory (SDT). Research shows SDT based treatment approaches can support engagement of intrinsic motivation and longterm integration of behavioural change. ADHD research shows individuals are impaired in some contexts but not in others and can manage well, indicating potential for ADHD neurodiverse "strengths" which could be developed and supported. Recent psychology research recommends cultivating positive psychological factors and emotions to improve mental health and wellbeing. Adults aged 18+ with a confirmed ADHD diagnosis will be invited to participate in two projects: Intensive online interviews of 1 hour will be conducted to identify, explore, and construct a theory about the factors, or "natural strengths" in lived experience of ADHD that help individuals to overcome everyday impairments. These factors will be incorporated into a pilot feasibility study of an SDT based 12-week treatment programme focusing on understanding the lived experience of ADHD and building on these strengths. The treatment will be designed for individual participants and delivered online. This study will have two sets of participants: one group will go directly to treatment, the other will go on a 12-week waiting list to create a comparison group. The second group will then be offered the 12-week treatment. Measures of experience of the participants will be looking for the feasibility, acceptability and efficacy of this treatment, as well as indicators of symptom improvement, and changes in self-awareness and self-regulation skills.

DETAILED DESCRIPTION:
ADHD symptoms negatively affect daily functioning both at work and at home, and have long-term impact in academic, occupational, social and emotional areas of functioning. Effective, long-term treatment outcomes benefit both the individual with ADHD and society as undiagnosed and untreated adults with ADHD may become an economic burden due to increased health care costs and decreased productivity at work. Russell Barkley postulated the first unifying theory of ADHD which places a core deficit of behavioural inhibition at the source of ADHD behaviours. Barkley's model is built upon observation of perceived chronic difficulties in behaviour, measured as "excessive or inappropriate for their age or development level.". Since the publication of this model, several theoretical models were proposed which attribute alternative cognitive sources for the development of ADHD symptoms, but Barkley's model forms the foundation for primary treatment recommendations. A recent review of the theories of ADHD recommended that more testable hypotheses need to be produced. While a variety of different interventions are available and the benefit of other forms of support is acknowledged (e.g. psychotherapy or coaching), the National Institute for Health and Care Excellence (NICE) only recommends interventions that match a similar protocol to medications: Randomised Controlled Trials (RCTs), which are primarily based in Cognitive Behavioural Therapy (CBT). It is therefore hypothesised that much of current research for the characterisation of ADHD is based on a cognitive behavioural paradigm that is deficit-focused with primary treatment outcomes of symptom reduction and control of maladaptive behaviours. Research in psychology suggests that a deficit-focus may not be the best approach to improving mental health, and it may be necessary to develop positive psychological factors and emotions that cultivate health and wellbeing. In ADHD, research suggests that this includes cognitive dynamism, creativity, and resilience, among others. There is a paucity of research in this area.

This project proposes an alternative approach to understanding and working with ADHD behaviours, supported by Self Determination Theory (SDT). SDT is an empirical, organismic dialectical approach to human motivation and personality, originating in Positive Psychology. SDT guided research focuses on conditions that enhance intrinsic motivation, self-regulation, and wellbeing. The positive approach to active energisation and intention of behaviour in SDT is closely aligned to evidence of positive engagement in ADHD (e.g. via interest), therefore viewing ADHD behaviours from an SDT perspective allows for a different understanding of the action and intention of behaviour. An SDT based approach combined with psychotherapeutic principles for integration of a positive concept of self provides tools which are potentially effective for long term treatment.

One of the challenges to designing effective treatment is the variability of impairment experienced by individuals with ADHD. Impairments are viewed as "clusters" of chronic difficulty for everyone with an ADHD diagnosis, however individual profiles can differ significantly. This implies there are situations or contexts where individuals with ADHD can function successfully. Two phases of this project have been developed to support this hypothesis. The aim of Phase 2 is to generate a theory, grounded in data, that explains a) why and how individuals with ADHD experience variable impairment; b) the impact of variable impairment for those with ADHD; and c) processes and strategies used by those with ADHD to resolve their main concerns regarding the impact and consequences of the variable impairment of ADHD. The purpose is to identify universal selective strengths that support individuals with ADHD to manage the variability of their impairment. In support of these alternative theories and approaches, Phase 3 of this project aims to examine the participant acceptability, feasibility, and efficacy of a novel strength - based programme of therapeutic self-development, psychoeducation and skills training for adults with a diagnosis of ADHD. This programme will use a multi-modal psychotherapeutic approach and educational methodology to assist participants in understanding ADHD and develop self-management skills.

While ADHD is primarily viewed as a neurobiological disorder with no cure, the possibility that ADHD may confer advantages to the individual is widely debated. Research on phenomena concerning the experience of ADHD has theoretical implications, and grounded theory is presented as a research methodology that is ideal for an area where not much research or theorising has been done before. There are currently several methodological approaches to grounded theory, and for this project it was deemed most appropriate to use a Constructivist approach. This approach introduces a pragmatic epistemological perspective on the researcher by recognising the subjectivity and researcher involvement in construction and interpretation of data in theory construction. This was thought to be an important element to monitor during the research process due to the researcher's own personal experience of ADHD.

In keeping with the focus on selecting cases which may provide new insights for developing theory, this project will aim to approach three different groups for participation: NHS patients from the Adult ADHD Clinic at the Southwest Yorkshire Partnership NHS Foundation Trust; university students at the University of Huddersfield and the University of Cambridge; and ADHD Support Groups for adults with ADHD. Analysis of individual case studies was considered, however as current perspectives of positive psychological factors in ADHD are identified as "individual strengths", it was thought a case comparison on interviews might identify the phenomenon in a more universal way.

The Phase 2 grounded theory research aims to reach saturation following analysis of 5-10 participant interviews. However, due to the nature of grounded theory, this can only be finalised as part of the process. It is possible more participants will

Unlike other qualitative methods, grounded theory approaches recommend that the inquiry shapes the data collection. This process of finding and generating data that is "rich", or detailed, focused, and full, provides solid material for substantive analysis. Therefore, this project will identify some areas to begin initial data collection, while remaining open to emerging potential data examples. These areas are intensive interviews, videos, and memos or field notes by the researcher.

Study Design - Pilot Study This is a wait list control study design with pre-, within, and post-treatment measures. A rolling entry of participants will be conducted, where once individuals have been screened their entry into the study will begin. A maximum of 30 adults aged 18+ with a confirmed diagnosis of ADHD will be allocated using block randomisation to the SDT theory-based model or wait list over a 12-week period. Following the 12-week wait, the wait list group will also be enrolled in the SDT theory-based model. This ensures all participants receive the opportunity to experience the treatment.

Participants will be recruited from NHS patients at the Adult ADHD Clinic at the Southwest Yorkshire Partnership NHS Foundation Trust only.Phase 3 is a pilot feasibility study, and the aim is to recruit 15 participants per arm for the two arm pilot study.

Acceptability, feasibility, and efficacy of the intervention will be measured by attendance and completion of evaluation forms at the end of each session. A follow up interview a week post-treatment will provide an opportunity for feedback and evaluation by post-treatment measures. Due to Covid-19 restrictions for research that requires in-person contact, consideration for the safety of participants and institution and NHS staff was incorporated into this study design. All interviews, screening, and treatment sessions will be conducted online, on an NHS approved video platform.

To test for treatment effects within the two groups, the psychometric data before and after therapy will be analysed statistically using a paired samples t-test, or dependant t-test. To test for treatment effects within the two groups, the psychometric data before and after therapy will be analysed statistically using the non-parametric paired-Wilcoxon test. Cohen's D will be calculated as a measure of effect size. To reduce bias, an intention to treat analysis will be used but it is recognised that challenges may occur due to missing data; based on withdrawal, loss to follow up, or non-response of assessment questionnaires and the degree of this this will be considered at the time of analysis. Therefore, the study will be reviewed using the revised Cochrane risk-of-bias tool for randomised trials (RoB 2). All analysis will be conducted with SPSS version 26.

The ethical process for this project is being reviewed by the University of Huddersfield School of Human and Health Sciences - School Research Ethics and Integrity Committee (SREIC) and will be reviewed by a relevant NHS ethics committee. Governance approvals will be obtained from university and NHS Trust sites. All sessions with Participants will be held in adherence with the Ethical Framework for Good Practice set by the UK Council for Psychotherapy (UKCP).

A British Association for Counselling and Psychotherapy (BACP) accredited psychotherapy supervisor will be engaged for two hours per month or one hour for every six patient sessions for the duration of the project to measure progress and review case work with participants if needed.

Participants will receive an invitation to an initial interview to discuss participation in the study. An information sheet detailing the purpose, activities, outcomes, and results of Phase 2 will be provided, including the researcher contact details (name, phone number, email address). Participants will be encouraged to read the information sheet again and ask questions on the assessment day prior to signing the consent form. The voluntary nature of participation and the ability to withdraw an individual's consent at any time will be emphasised during the study.

For the Phase 2 intensive interviews, all participants will be entered into a draw for a £50 Amazon voucher. This was suggested by the lived experience group as contribution to research for ADHD was not considered enough of a benefit alone.

For participants in the Phase 3 pilot study, they will receive 11 weekly sessions of individually focused therapeutic coaching support which is not currently accessible within the service. It is possible that a waitlist control design study might be an incentive for participants to join, as all participants in the study will eventually receive the intervention. However, we considered it unethical to offer a place in the study without the option to receive the intervention. Participants will be given a minimum of 24 hours and up to three days to consider participation in the study, and the researcher will be available to answer any questions they have.

A critical element of this research project is the exploration and representation of the lived experience of adults with ADHD, and the applicability, efficacy, and accessibility of the results. Therefore, this project has involved a patient participation group in pre-study preparation before recruitment. A small group of 5-6 adults with ADHD who expressed strong interest in the research have reviewed and refined recruitment materials for Phase 2 and Phase 3, including the recruitment flyers, patient information sheets, consent forms and interview guide.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of ADHD
* Age 18 or older
* Access to computer or smartphone with an internet connection

Exclusion Criteria:

* Co-morbid diagnosis (e.g. Autism, Bi-polar, Learning Disabilities, Traumatic Brain Injury, Psychosis or Tourette's)
* Substance abuse disorders
* Other mental health disorders (e.g. PTSD, Oppositional Defiant Disorder
* Personality Disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Weiss Functional Impairment Rating Scale -WFIRS | Baseline and immediately after intervention
  Measures change in severity of ADHD symptoms. Lilkert scale where the total score can be reviewed, or a mean score from each relevant domain. Higher scores mean worse outcome.
Patient Heath Questionniare (PHQ)- 9 | Baseline and immediately after intervention
  Major Depressive Disorder section of larger PHQ measuring change in severity of Depression symptoms. Minimim score 0, maximum score 27, higher scores mean worse outcome.
General Anxiety Disorder (GAD) 7 | Baseline and immediately after intervention
  Measures change in severity of Anxiety symptoms. Scale score ranges from 0 to 21 with cut points of 5, 10, and 15 that might be interpreted as representing mild, moderate, and severe levels of anxiety. Higher scores mean worse outcome.
Harter's Self Perception Profile | Baseline and immediately after intervention
  Measures changes in self awareness. Each item has minimum score of 1, maximum score of 4. Mean scores are calculated for each of 12 sub-domains. Higher scores mean better outcome.
Index of Autonomous Functioning -IAF | Baseline and immediately after intervention
  Measures changes in feeling self-determined. Each item scores minimum 1, maximum 5 and total is calculated by averaging scores from 15 items. Higher scores mean better outcome.
Perceived Choice and Awareness of Self Scale -PCASS | Baseline and immediately after intervention
  Measures changes in feeling self-determined. Likert 10-item scale, with two 5-item subscales with minimum of 1 and maximum of 5 on each item. Total is calculated by averaging scores in each subscale, with higher scores meaning a better outcome.
Personal Questionnaire - PQ | During the intervention
  Measure change in participant selected specific psychological difficulties. 10 problems are measured weekly with score of minimum 1, maximum 7. Total is calculated by averaging scores in each subscale, with higher scores meaning a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Tolchard, Study Chair — University of Huddersfield
Locations (2):
- United Kingdom (2):
  - University of Huddersfield, Huddersfield, West Yorkshire
  - Manygates Adult ADHD Clinic, Wakefield, West Yorkshire

IPD SHARING:
Plan to Share IPD: No
To protect identity of individual participants, all personally identifiable data (PID) will be anonymised and will not be released. All participant case records will be held in accordance with the Data Protection Act. Records will be kept both in electronic and hard copy form. The participants' home addresses and telephone numbers will be kept on a secure database and spreadsheet on NHS/University computers in compliance to the Data Protection Act. Data held in the NVivo database will be anonymised and only accessible by password protected researcher login. All manual records will be kept in a locked cabinet accessible by the researcher only.
  In accordance with the Data Protection Act personal data will not be retained for longer than is necessary. The University of Huddersfield recommends that data is stored for 10 years to aid transparency and integrity of research. Long term storage of data will be accessible by the researcher only.

REFERENCES:
- [Background] Armstrong, T. (2010). The Power of Neurodiversity: Unleashing the Advantages of Your Differently Wired Brain. Philadelphia, PA: Da Capo Press.
- [Background] Barkley RA. Behavioral inhibition, sustained attention, and executive functions: constructing a unifying theory of ADHD. Psychol Bull. 1997 Jan;121(1):65-94. doi: 10.1037/0033-2909.121.1.65. PMID 9000892
- [Background] Barkley RA. Major life activity and health outcomes associated with attention-deficit/hyperactivity disorder. J Clin Psychiatry. 2002;63 Suppl 12:10-5. PMID 12562056
- [Background] Barkley, R. (2012). Executive Functions: What They Are, How They Work, and Why They Evolved. New York, NY: Guildford Press.
- [Background] Bazeley, P. (2007). Qualitative Data Analysis with NVivo. London: SAGE Publications Ltd.
- [Background] Bokor G, Anderson PD. Attention-Deficit/Hyperactivity Disorder. J Pharm Pract. 2014 Aug;27(4):336-49. doi: 10.1177/0897190014543628. PMID 25092688
- [Background] Boot, N. (2017). The creative brain: Subclinical Symptoms of Attention-Deficit/Hyperactivity Disorder (ADHD) are Associated with Specific Creative Processes. In The Creative Brain (pp. 71-98). UvA-DARE (Digital Academic Repository)
- [Background] Bringer, J. D., Johnston, L. H., & Brackenridge, C. H. (2004). Maximising transparancy in a doctoral thesis: the complexities of writing about the use of QSR*NVIVO within a grounded theory study. Qualitative Research, 4(2), 247-265
- [Background] Brooks, R. B. (2002). Changing the Mindset of Adults with ADHD: Strategies for Fostering Hope, Optimism, and Resilience. In S. Goldstein & A. T. Ellison (Eds.), Clinician's guide to adult ADHD: Assessment and intervention (pp. 127-146). San Diego, CA: Academic Press
- [Background] Brown TE. ADD/ADHD and Impaired Executive Function in Clinical Practice. Curr Psychiatry Rep. 2008 Oct;10(5):407-11. doi: 10.1007/s11920-008-0065-7. PMID 18803914
- [Background] Canu WH, Hartung CM, Stevens AE, Lefler EK. Psychometric Properties of the Weiss Functional Impairment Rating Scale: Evidence for Utility in Research, Assessment, and Treatment of ADHD in Emerging Adults. J Atten Disord. 2020 Oct;24(12):1648-1660. doi: 10.1177/1087054716661421. Epub 2016 Aug 1. PMID 27481918
- [Background] Charmaz, K. (2014). Constructing Grounded Theory. London: SAGE Publications Ltd.
- [Background] Deci, E., & Ryan, R. (1985). Intrinsic Motivation and Self Determination in Human Behaviour. New York: Plenum Press.
- [Background] Flick, U. (2018a). An Introduction to Qualitative Research. London: SAGE Publications Ltd.
- [Background] Flick, U. (2018b). Doing Grounded Theory. London: SAGE Publications Ltd
- [Background] Fullen, T., Jones, S. L., Marie, L., & Adamou, M. (2020). Psychological Treatments in Adult ADHD: A Systematic Review. Journal of Psychopathology and Behavioural Assessment.
- [Background] Gawler-Wright, P., & Rossi, E. (2013). Introduction to the Principles of Contemporary Psychotherapy. London: Beeleaf Publishing.
- [Background] Gibbs, G. (2018). Analysing Qualitative Data. London: SAGE Publications Ltd.
- [Background] Glaser, B. (1978). Theoretical sensitivity. Mill Valley, California: Sociology Press.
- [Background] Glaser, B. (1992). Basics of Grounded Theory Analysis: Emergence Vs. Forcing. Mill Valley, California: Sociology Press.
- [Background] Glaser, B., & Strauss, A. (1967). The Discovery of Grounded Theory: Strategies for Qualitative Research. New York, NY: Routledge
- [Background] Great Britain: Parliment. (1998). Data Protection Act. Retrieved 29 December 2014, from http://www.legislation.gov.uk/ukpga/1998/29/contents
- [Background] Hartmann, T. (1997). ADD: A Different Perception. Grass Valley, California: Underwood Books.
- [Background] Hutchison, A. J., Johnston, L. H., Breckon, J. D., John, A., Johnston, L. H., & Breckon, J. D. (2010). Using QSR - NVivo to facilitate the development of a grounded theory project : an account of a worked example. International Journal of Social Research Methodology, 13(4), 283-302.
- [Background] Jacob KS. Recovery model of mental illness: a complementary approach to psychiatric care. Indian J Psychol Med. 2015 Apr-Jun;37(2):117-9. doi: 10.4103/0253-7176.155605. No abstract available. PMID 25969592
- [Background] Johnson KA, Wiersema JR, Kuntsi J. What would Karl Popper say? Are current psychological theories of ADHD falsifiable? Behav Brain Funct. 2009 Mar 3;5:15. doi: 10.1186/1744-9081-5-15. PMID 19257888
- [Background] Kooij JJS, Bijlenga D, Salerno L, Jaeschke R, Bitter I, Balazs J, Thome J, Dom G, Kasper S, Nunes Filipe C, Stes S, Mohr P, Leppamaki S, Casas M, Bobes J, Mccarthy JM, Richarte V, Kjems Philipsen A, Pehlivanidis A, Niemela A, Styr B, Semerci B, Bolea-Alamanac B, Edvinsson D, Baeyens D, Wynchank D, Sobanski E, Philipsen A, McNicholas F, Caci H, Mihailescu I, Manor I, Dobrescu I, Saito T, Krause J, Fayyad J, Ramos-Quiroga JA, Foeken K, Rad F, Adamou M, Ohlmeier M, Fitzgerald M, Gill M, Lensing M, Motavalli Mukaddes N, Brudkiewicz P, Gustafsson P, Tani P, Oswald P, Carpentier PJ, De Rossi P, Delorme R, Markovska Simoska S, Pallanti S, Young S, Bejerot S, Lehtonen T, Kustow J, Muller-Sedgwick U, Hirvikoski T, Pironti V, Ginsberg Y, Felegyhazy Z, Garcia-Portilla MP, Asherson P. Updated European Consensus Statement on diagnosis and treatment of adult ADHD. Eur Psychiatry. 2019 Feb;56:14-34. doi: 10.1016/j.eurpsy.2018.11.001. Epub 2018 Nov 16. PMID 30453134
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Kuntsi J, Klein C. Intraindividual variability in ADHD and its implications for research of causal links. Curr Top Behav Neurosci. 2012;9:67-91. doi: 10.1007/7854_2011_145. PMID 21769722
- [Background] Lempert, L. B. (2007). 'Asking Questions of the data: memo writing in the grounded theory tradition'. In A. Bryant & K. Charmaz (Eds.), The SAGE Handbook of Grounded Theory (pp. 245-265). London: SAGE Publications Ltd.
- [Background] Liberman, R. P. (2008). Recovery from disability: Manual of psychiatric rehabilitation. Arlington, VA: American Psychiatric Publishing, Inc..
- [Background] Messer, B., & Harter, S. (2012). The Self-Perception Profile for Adults: Manual and Questionnaires. Denver, Colorado: University of Denver.
- [Background] Morse, J. M. (1998). 'Designing funded qualitative research'. In N. Denzin & Y. Lincoln (Eds.), Strategies of Qualitative Inquiry (pp. 56-85). London: SAGE Publications Ltd
- [Background] Newark PE, Stieglitz RD. Therapy-relevant factors in adult ADHD from a cognitive behavioural perspective. Atten Defic Hyperact Disord. 2010 Jun;2(2):59-72. doi: 10.1007/s12402-010-0023-1. Epub 2010 Apr 15. PMID 21432591
- [Background] Attention deficit hyperactivity disorder: diagnosis and management. London: National Institute for Health and Care Excellence (NICE); 2019 Sep. Available from http://www.ncbi.nlm.nih.gov/books/NBK493361/ PMID 29634174
- [Background] Nimmo-Smith V, Merwood A, Hank D, Brandling J, Greenwood R, Skinner L, Law S, Patel V, Rai D. Non-pharmacological interventions for adult ADHD: a systematic review. Psychol Med. 2020 Mar;50(4):529-541. doi: 10.1017/S0033291720000069. Epub 2020 Feb 10. PMID 32036811
- [Background] Philipsen A, Richter H, Peters J, Alm B, Sobanski E, Colla M, Munzebrock M, Scheel C, Jacob C, Perlov E, Tebartz van Elst L, Hesslinger B. Structured group psychotherapy in adults with attention deficit hyperactivity disorder: results of an open multicentre study. J Nerv Ment Dis. 2007 Dec;195(12):1013-9. doi: 10.1097/NMD.0b013e31815c088b. PMID 18091195
- [Background] Ramsay, J. R. (2010). CBT for Adult ADHD: Adaptations and Hypothesized Mechanisms of Change. Journal of Cognitive Psychotherapy, 24(1), 37-45
- [Background] Ramsay, J. R., & Rostain, A. L. (2015). The Adult ADHD Toolkit. New York: Routledge
- [Background] Richards, L. (2002). Qualitative computing--a methods revolution? International Journal of Social Research Methodology, 5(3), 263-276
- [Background] Roberts, W., Milich, R., & Barkley, R. (2014). Primary Symptoms, Diagnostic Criteria, Subtyping and Prevalence of ADHD. In R. Barkley (Ed.), Attention Deficit Hyperactivity Disorder: A Handbook for Diagnosis and Treatment (4th ed., pp. 51-80). New York: Guilford Press.
- [Background] Rogers, C. (1951). Client-centered therapy: Its current practice, implications and theory. Boston, MA: Houghton Mifflin.
- [Background] Rostain AL, Ramsay JR. A combined treatment approach for adults with ADHD--results of an open study of 43 patients. J Atten Disord. 2006 Nov;10(2):150-9. doi: 10.1177/1087054706288110. PMID 17085625
- [Background] Ryan RM, Deci EL. Self-determination theory and the facilitation of intrinsic motivation, social development, and well-being. Am Psychol. 2000 Jan;55(1):68-78. doi: 10.1037//0003-066x.55.1.68. PMID 11392867
- [Background] Ryan, Richard, & Deci, E. (2017). Self-Determination Theory Basic Psychological Needs in Motivation, Development, and Wellness. New York, NY: Guilford Press.
- [Background] Ryan RM, Deci EL. Intrinsic and Extrinsic Motivations: Classic Definitions and New Directions. Contemp Educ Psychol. 2000 Jan;25(1):54-67. doi: 10.1006/ceps.1999.1020. PMID 10620381
- [Background] Safren, S., Perlman, C., Sprich, S., & Otto, M. (2005). Mastering Your Adult ADHD. New York: Oxford University Press.
- [Background] Sagvolden T, Johansen EB, Aase H, Russell VA. A dynamic developmental theory of attention-deficit/hyperactivity disorder (ADHD) predominantly hyperactive/impulsive and combined subtypes. Behav Brain Sci. 2005 Jun;28(3):397-419; discussion 419-68. doi: 10.1017/S0140525X05000075. PMID 16209748
- [Background] Sedgwick JA, Merwood A, Asherson P. The positive aspects of attention deficit hyperactivity disorder: a qualitative investigation of successful adults with ADHD. Atten Defic Hyperact Disord. 2019 Sep;11(3):241-253. doi: 10.1007/s12402-018-0277-6. Epub 2018 Oct 29. PMID 30374709
- [Background] Sergeant J. The cognitive-energetic model: an empirical approach to attention-deficit hyperactivity disorder. Neurosci Biobehav Rev. 2000 Jan;24(1):7-12. doi: 10.1016/s0149-7634(99)00060-3. PMID 10654654
- [Background] Shaw M, Hodgkins P, Caci H, Young S, Kahle J, Woods AG, Arnold LE. A systematic review and analysis of long-term outcomes in attention deficit hyperactivity disorder: effects of treatment and non-treatment. BMC Med. 2012 Sep 4;10:99. doi: 10.1186/1741-7015-10-99. PMID 22947230
- [Background] Sheldon, K. M., & Ryan, R. M. (1996). Percieved Choice and Awareness of Self Scale (PCASS), University of Rochester
- [Background] Solanto, M. V. (2010). Cognitive-Behavioural Therapy for Adult ADHD. New York: Guildford Press.
- [Background] Solanto MV, Marks DJ, Mitchell KJ, Wasserstein J, Kofman MD. Development of a new psychosocial treatment for adult ADHD. J Atten Disord. 2008 May;11(6):728-36. doi: 10.1177/1087054707305100. Epub 2007 Aug 21. PMID 17712167
- [Background] Sonuga-Barke EJ. Psychological heterogeneity in AD/HD--a dual pathway model of behaviour and cognition. Behav Brain Res. 2002 Mar 10;130(1-2):29-36. doi: 10.1016/s0166-4328(01)00432-6. PMID 11864715
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Stein DJ, Fan J, Fossella J, Russell VA. Inattention and hyperactivity-impulsivity: psychobiological and evolutionary underpinnings of ADHD. CNS Spectr. 2007 Mar;12(3):190, 193-6. doi: 10.1017/s1092852900020903. PMID 17329979
- [Background] Strauss, A., & Corbin, J. (1998). Basics of Qualitative Research: Grounded Theory Procedures and Techniques. London: SAGE Publications Ltd.
- [Background] UK Council for Psychotherapy. (2019). UKCP Code of Ethics and Professional Practice. London: UK Council for Psychotherapy.
- [Background] Wake, L. (2008). Neurolinguistic Psychotherapy: A Postmodern Perspective. New York: Routledge.
- [Background] Walter, J. G., & Hart, J. (2009). Understanding the complexities of student motivations in mathematics learning. Journal of Mathematical Behavior, 28(2-3), 162-170.
- [Background] Weinstein, N., Przybylski, A. K., & Ryan, R. M. (2012). The index of autonomous functioning: Development of a scale of human autonomy. Journal of Research in Personality, 46(4), 397-413.
- [Background] Weiss M, Murray C, Wasdell M, Greenfield B, Giles L, Hechtman L. A randomized controlled trial of CBT therapy for adults with ADHD with and without medication. BMC Psychiatry. 2012 Apr 5;12:30. doi: 10.1186/1471-244X-12-30. PMID 22480189
- [Background] White, H. A., & Shah, P. (2011). Creative style and achievement in adults with attention-deficit/hyperactivity disorder. Personality and Individual Differences, 50(5), 673-677.
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Young, S. (1999). Psychological therapy for adults with Attention Deficit Hyperactivity Disorder. Counselling Psychology Quarterly, 12(2), 183-190.
- [Derived] Champ RE, Meneses RW, Adamou M, Gillibrand W, Arrey S, Tolchard B. A Neuroaffirmative, Self-Determination Theory-Based Psychosocial Intervention for Adults With Attention-Deficit/Hyperactivity Disorder: Randomized Feasibility Study. JMIR Form Res. 2025 Oct 29;9:e69943. doi: 10.2196/69943. PMID 41161339